CLINICAL TRIAL: NCT02495740
Title: E-Bike Study - Endurance Capacity Following 1 Month Training of Classic Bike Versus Electric-assisted Bike
Brief Title: E-Bike Versus Classic Bike Intervention Trial
Acronym: E-bike
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Arno Schmidt-Trucksäss, Prof. Dr. Arno Schmidt-Trucksäss, University of Basel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EKNZ 2012/164
Record Dates: First submitted 2015-07-09; First posted 2015-07-13 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Physical Activity; Obesity
MeSH Terms: conditions — Motor Activity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- E-bike intervention (Experimental): Intervention is active commuting to work by an electric assisted bike to work for a period of 4 weeks at least 3 times per week with a minimal distance of 6 km per way
  Interventions: Behavioral: Commuting to work
- Bike intervention (Active Comparator): Intervention is active commuting to work by classic bike for a period of 4 weeks at least 3 times per week with a minimal distance of 6 km per way
  Interventions: Behavioral: Commuting to work

INTERVENTIONS:
Behavioral: Commuting to work — Commuting by an electric assisted bike to work for a period of 4 weeks at least 3 times per week

SUMMARY:
The effects of active commuting with an e-bike, as compared with a "classic" bike, on cardiorespiratory fitness and vascular health are largely unknown. To assess whether active commuting with an e-bike or a classic bike increases peak oxygen consumption (VO2peak) in untrained and overweight individuals.

DETAILED DESCRIPTION:
Riding an electrically assisted bicycle (e-bike) is thought to be suitable to increase physical activity in daily life, to promote health, and to increase cardiorespiratory fitness in normal-weight individuals. The positive effect of commuting to work by a normal bike on cardiorespiratory fitness has been shown to be an important predictor of cardiovascular mortality in previous studies. We thought to improve maximal oxygen uptake by commuting to work by e-bike vs. classic bike. Besides cardiorespiratory fitness we assessed arterial stiffness as brachial-ankle pulse wave velocity as an independent predictor of cardiovascular events and all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

body mass index 25-35 kg/m2, and willingness to commute to work by e-bike or by normal bike at least 3 times per week with a one-way distance of ≥ 6 km.

Exclusion Criteria:

cycling as a leisure-time activity, active commuting to work or exercise training more than once per week within 4 weeks before the start of the study, uncontrolled cardiovascular diseases limiting cardiorespiratory fitness, stage II arterial hypertension (systolic blood pressure > 160 mmHg, diastolic blood pressure > 95 mmHg), renal diseases, uncontrolled diabetes mellitus (HbA1c > 6.5%), or active malignancy or chemotherapy during the past 6 months.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
maximal oxygen uptake | 4 weeks
  maximal oxygen uptake measured on a cycle ergometer with a ramp protocol

CONTACTS AND LOCATIONS:
Overall Officials: Arno Schmidt-Trucksäss, Principal Investigator — University of Basel
Locations (1):
- Department for Sport, Exercise and Health, Sports and Exercise Medicine, University of Basel, Basel, Switzerland